CLINICAL TRIAL: NCT06331988
Title: Microbiome,Immune-system and Tumor Interaction in Colorectal Cancer (MITICO Study)
Brief Title: Microbiome, Immune-system and Tumor Interaction in Colorectal Cancer
Acronym: MITICO
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1341
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: microbioma; Immune-system; Colorectal Cancer; risk factor; micro-environmental factors
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, oral swab, faecal and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- resectable colorectal cancer patient: patients with resectable CRC candidate to radical surgery and - after approximately 4-8 weeks - adjuvant chemotherapy (if indicated), accordingly to standard of care (SOC)

SUMMARY:
Colorectal cancers represent the second leading cause of cancer-related death in the United States Western world. In Italy they represent the second most frequent neoplasm (49,000 cases in 2019). Despite the advancement of surgical techniques and medical therapy programs systemic, it is estimated that approximately 40-50% of colorectal cancers recur after being treated for a limited loco-regional disease. Patients who develop metastases throughout their history clinic have a 5-year overall survival of just over 10%.

Adjuvant systemic chemotherapy can reduce the risk of disease recurrence in patients with colorectal adenocarcinomas, however, the standard drugs used to date for this use (fluoropyrimidines and oxaliplatin) have not undergone substantial changes in the last 20 years or so.

A crucial point is the need to have more precise information regarding risk factors above all biomolecular to base therapeutic choices.

It has now become urgent to overcome the T-tumor N-node M- metastasis (TNM) staging, to have more modern knowledge on the factors capable of impacting significantly on the prognosis, influence the real risk of disease recurrence, Identify new prognostic categories and subcategories, therefore being able to predict the clinical benefit of treatments that can be more targeted, personalized and effective. In this panorama it has developed in recent years an ever-growing literature also regarding the role of bacterial flora intestinal (microbiota) in patients with colorectal cancer. In particular, recent discoveries have highlighted the immunoregulatory role of the microbiota in the anti-tumor response. This study aims of evaluating how the molecular characteristics of the tumor, of the infiltrating immune system cells and of the associated intestinal microbiota correlate with the development of colorectal cancer, its progression and response to treatments.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related mortality. Despite the improvement of surgical techniques, ~30-50% of patients with locoregional CRC who undergo potentially curative surgery ultimately relapse and die of metastatic disease. On the other hand, it is also well established that adjuvant systemic chemotherapy can decrease the risk of death in these patients.

Currently, the standard treatment of locoregional CRC is based on curative surgery alone or followed by adjuvant systemic chemotherapy based on risk factors. In this regard, international guidelines recommend chemotherapy for stage III and stage II colon cancer with high risk prognostic characteristics, including T4 lesions, poorly differentiated tumors, lymphovascular or perineural invasion, tumour presentation with obstruction or tumour perforation, positive margins, and inadequate (<12) number of lymph nodes analyzed after surgery. In patients treated with surgery and adjuvant systemic chemotherapy the 3-year disease-free survival (3y DFS) is 72% in stage III patients and 87% in stage II patients.The risk factors known to date do not always correctly predict the prognosis in these patients. For example, tumors of the same stage can largely differ in both prognosis, which can lead to wrong treatment decisions. This means that our knowledge about factors influencing the chance of recurrence and the prediction of benefit from systemic treatment is limited. Identification of these factors along with better treatment strategies may help in reducing the recurrence rate and raising the life expectancy of CRC patients. In this regard, the role of commensal microbiota in CRC development and response to treatments is emerging as a critical factor. The term microbiome "refers to the microorganisms involved but also encompasses their theatre of activity". In a mutually beneficial and dynamic equilibrium, bacteria coexist on our body stimulating the basal production of tissue repair factors while immune system surveils on pathogens outgrowth. The gut microbiota has been consistently shown to play a role in the development of CRC, The present project will establish the foundation of methods for early detection of the microbiome-immune-induced mutator phenotypes involved in the relapse. Results from this study will pave the way for future interventions to constrain the mutation rates of tumor.

Through this prospective observational Microbiome Immune-system Tumor Interaction in Colorectal Oncology (MITICO) project a new platform will be established integrating patient's clinical and lifestyle information with genomic data from both, CRC and the commensal microbiota, along with profiling of local and systemic immune responses.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years of age
* Histologically proven adenocarcinoma of the colon and superior rectal cancer suitable for primary curative surgery at European Oncology Institute and followed by adjuvant chemotherapy if indicated.
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0-1
* Written informed consent
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and all protocol procedures.

Exclusion Criteria:

* Evidence of metastatic colon cancer at diagnosis
* Previous or concurrent malignancies, except for adequately treated basal or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years prior to study entry
* Psychiatric disorder precluding understanding of information on trial-related topics or giving informed consent or interfering with compliance for treatment schedule
* Any serious underlying medical conditions or serious co-morbidities which could impair the prognosis and/or the ability of the patient to participate in this trial
* Patients with active autoimmune diseases such as Inflammatory Bowel Disease, Lupus, etc. or other conditions requiring systemic corticosteroids or other systemic immunosuppressive medications.
* Use of antibiotics within 45 days from the enrollment.
* Pregnant or lactating females.
* Unwillingness or inability to follow the procedures required in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resectable CRC candidate to radical surgery and - after approximately 4-8 weeks - adjuvant chemotherapy (if indicated), accordingly to standard of care (SOC).
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 5 years
  To define the association between mucosal microbiota and 3y DFS in CRC patients underwent surgical resection +/- adjuvant chemotherapy

SECONDARY OUTCOMES:
Overall survival | 5 years
  To define the association between faecal microbiota and 3-year disease free survival (3y DFS) and 5y Overall survival (OS). To define the association between tumor intrinsic and extrinsic features and:
  * 3y DFS -5y OS
  * Tumor localization (e.g. right versus left)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Ciardiello, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No